CLINICAL TRIAL: NCT07133737
Title: Follow-up Study of at Least 5 Years After a SMILE® Pro Procedure for the Correction of Hyperopia Investigating Long-term Visual Outcomes and Potential Side Effects
Brief Title: 5 Year Follow up of SMILE® Procedure for the Correction of Hyperopia
Acronym: PHOBOS-5FU
Status: Enrolling by invitation | Type: Observational
Sponsor: Gemini Eye Clinic (Industry)
Responsible Party: Principal Investigator, Dr. Pavel Stodulka, Principal Investigator, Gemini Eye Clinic
Other Study IDs: PHOBOS-5FU
Record Dates: First submitted 2025-08-08; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Hyperopia
Keywords: relex; smile; eye surgery; hyperopia
MeSH Terms: conditions — Hyperopia; Smiling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- post hyperopia correction: Patients who underwent hyperopia correction surgery using Femtosecond laser system VisuMax with treatment option ReLEx SMILE at least 5 years ago and were part of the original clinical investigation

SUMMARY:
The planned study will investigate and evaluate refractive stability, predictability, and safety in patients who underwent SMILE® pro surgery for hyperopia with or without astigmatism at least five years ago.

This study aims to gain long-term insights into the predictability, safety, stability and side effects of the SMILE® pro procedure. It will evaluate the refractive outcome so the findings can optimize treatment nomograms and selection criteria while providing evidence of the long-term stability and predictability of the procedure.

Approximately 100 patients in the Czech Republic and Germany will participate in this study. The study was reviewed and approved by an independent research ethics committee.The study will consist of a single visit, where standard, non-invasive and painless examinations will be performed. The course of this visit will correspond to the patient's last visit five years ago as part of the clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent the SMILE hyperopic procedure as part of the study referenced PHOBOS.
* Patients should be able to understand the patient information and willing to sign an informed consent.
* Patients should be willing to comply with all examinations during the visit.

Exclusion Criteria:

* Patients with severe ocular or generic disorders that would prevent them from completed the visit.
* Patients not being able to understand and give informed consent.
* Patients who did not underwent the SMILE hyperopic procedure as part of the study referenced PHOBOS.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population are patients who suffered from hyperopia and hyperopia with astigmatism (including presbyopic patients who might have a myopic target) and underwent the original PHOBOS clinical study are medically suitable to undertake the current clinical study investigation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Loss of more than 2 lines of CDVA | Baseline, 12 months, 5 years
  Less than 5.0% of eyes loose more than 2 lines of CDVA at 5 years follow-up compared to the baseline visit.
Manifest refractive astigmatism greater than 2.0 D | 5 years
  Induced manifest refractive astigmatism greater than 2.0 D should occur in less than 5% of subjects at 5 years follow-up.
MRSE stability within ±1.0 D | 12 months, 5 years
  At least 95% of eyes should be stable with a change in Manifest Refractive Spherical Equivalent within ±1D between 12 months and 5 years follow-up visits.
CDVA worse than 20/40 | 5 years
  Less than 1.0% of eyes have a post-operative CDVA worse than 20/40 at 5 years follow-up.
UDVA better than 20/40 | 5 years
  At least 85% of eyes intended for emmetropia achieve an UDVA of 20/40 or better at 5 years follow-up.
MRSE target within ±0.5 D | 5 years
  Post-operative SE relative to the intended target should be within ±0.50D in ≥50% of eyes.
MRSE target within ±1.0 D | 5 years
  Post-operative SE relative to the intended target should be within ±1.00 D ≥75% of eyes.

SECONDARY OUTCOMES:
Change in CDVA | Baseline, 12 months, 5 years
  Change in CDVA as a loss-of-line distribution at each time point (safety diagram)
Distribution of CDVA | Baseline, 12 months, 5 years
  Cumulative distribution of CDVA at each time point including safety index
Distribution of UDVA | Baseline, 12 months, 5 years
  Cumulative UDVA distribution at each time point compared to pre-operative CDVA
Distribution of UNVA | Baseline, 12 months, 5 years
  Cumulative UNVA distribution at each time point.
Distribution of MRSE | Baseline, 12 months, 5 years
  Spherical equivalent refractive accuracy
Change of MRSE | Baseline, 12 months, 5 years
  Stability of spherical equivalent refraction
Change of subjective refractive astigmatism | Baseline, 12 months, 5 years
  Stability of subjective refractive astigmatism
Adverse events incidence | Baseline, 12 months, 5 years
  Intraoperative and adverse events at each time point (numbers and percentages)
Quality of vision | 5 years
  Evaluation of patient satisfaction using patient questionnaire with focus on quality of vision. A Rasch-Analysis will be performed based on a questionnaire to evaluate the QoV (Quality of Vision) with a lower score indicating better vision and higher worse vision.
Contrast sensitivity changes | Baseline, 12 months, 5 years
  Determination of contrast sensitivity measured by CSV 1000 (Vector Vision) (changes from the pre-operative to the post-operative state and its stability over time will be investigated).
Change in corneal keratometry | Baseline, 12 months, 5 years
  Comparision of mean corneal keratometry with an analysis diameter of 6 mm.
Change in higher order corneal abberations | Baseline, 12 months, 5 years
  Comparision of higher order corneal abberations with an analysis diameter of 6 mm.
Corneal epithelium thickness | 5 years
  Analysis of corneal epithelium thickness with an analysis of min-max difference in a diameter of 6 mm.
Pentacam Nucleaus Staging | 5 years
  Rate of Pentacam Nuclear Staging (PNS) providing a cataract grading score on an ordinal scale (from 0 to 5) where 0 is no cataract.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Stodulka, Dr. Ph.D, FEBOS-CR, Principal Investigator — Gemini Eye Clinic; Anke Messerschmidt-Roth, Dr. rer. medic., Principal Investigator — Klinik für Augenheilkunde Marburg; Walter Sekundo, Prof. Dr. med., Principal Investigator — Klinik für Augenheilkunde Marburg
Locations (2):
- Gemini Eye Clinic, Zlín, Czechia
- Universitätsklinikum Marburg - Klinik für Augenheilkunde, Marburg, Germany

REFERENCES:
- [Background] Waring GO 3rd, Reinstein DZ, Dupps WJ Jr, Kohnen T, Mamalis N, Rosen ES, Koch DD, Obstbaum SA, Stulting RD. Standardized graphs and terms for refractive surgery results. J Refract Surg. 2011 Jan;27(1):7-9. doi: 10.3928/1081597X-20101116-01. No abstract available. PMID 21229953
- See also: the protocol of the original study - ClinicalTrials.gov ID: NCT03431571 — https://clinicaltrials.gov/study/NCT03431571?locStr=Czech%20Republic&country=Czechia&term=NCT03431571&rank=1